CLINICAL TRIAL: NCT03150043
Title: Continuous Non-Invasive Measurement of Hemoglobin During Parturition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-0087
Record Dates: First submitted 2017-05-08; First posted 2017-05-11 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2018-04

CONDITIONS: Hemorrhage; Cesarean Section
Keywords: Hemoglobin; Cesarean delivery
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: All patients who agree to participate in the study will have the non-invasive hemoglobin monitor placed on their finger during delivery. The values obtained from the non invasive monitor will be masked to the clinicians during delivery. No medical decision making will be based on values obtained from the non-invasive monitor. After the patient leaves the recovery room, values obtained from the monitor will be compared to those obtained via blood draw. Patients will be separated into quartiles based on drop in hemoglobin (between pre-op and post-op day 1) and hemoglobin values obtained from the monitor will be compared between the quartiles.
Masking Description: Since every patient will have the device placed during delivery, there will be no masking. However, the actual values obtained from the monitor will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All Participants (Other): All patients who agree to participate in the study will have the Masimo Rainbow Pulse CO-Oximeter non-invasive hemoglobin monitor placed on their finger during cesarean delivery. A CBC will be drawn immediately prior to delivery and this value will be compared to the values obtained from the monitor. The patients will be separated into quartiles based on total drop in hemoglobin (pre-op to post-op day 1) and the values from the monitor compared between quartiles.
  Interventions: Device: Masimo Rainbow Pulse CO-oximeter

INTERVENTIONS:
Device: Masimo Rainbow Pulse CO-oximeter — Masimo Rainbow Pulse CO-oximeter will be used to measure hemoglobin values of pregnant women during primary cesarean delivery

SUMMARY:
A non-invasive hemoglobin monitor will be used during cesarean delivery and the values obtained will be compared to values obtained from traditional blood draw.

DETAILED DESCRIPTION:
Obstetric hemorrhage remains the leading cause of maternal death worldwide (2). The most common culprits are uterine atony, placental disorders, and delivery trauma. Current detection and management of hemorrhage is heavily based on clinical judgment and laboratory results. Interventions such as fluid resuscitation and blood transfusion are often initiated after a significant hemorrhage has already taken place. Early detection and treatment of this potentially life threatening obstetric complication is of upmost importance in the field of obstetrics. Traditional methods for assessing hemoglobin levels involve collecting the patient's blood and sending it to the laboratory for analysis via complete blood count (CBC). This involves a delay and often patients are continuing to hemorrhage while the CBC is being processed. Novel technology has recently been approved by the FDA, which can continuously assess hemoglobin levels via a non-invasive monitor. This device works as a pulse oximeter, which is placed on the index finger and uses infrared technology to estimate hemoglobin levels (1). Despite its validation and use in many patient populations such as trauma, neurosurgery and orthopedic surgery, data is lacking in an obstetric population. The investigator's hypothesis is that this device will enable clinicians detect hemorrhage early and initiate resuscitation such as fluid and/or blood transfusion before significant hemorrhage has taken place. This study will be a proof of concept prospective cohort study, in which the investigators will attempt to detect the association between intra-operative and postoperative continuous non-invasive hemoglobin monitoring and postpartum decrease in hemoglobin.

Women undergoing primary cesarean delivery after failed induction of labor or repeat cesarean delivery after failed TOLAC (trial of labor after cesarean delivery), will be eligible for participation in this study. Prior to cesarean, all patients will have a CBC drawn. Masimo non-invasive hemoglobin monitor will be placed on their finger during delivery and remain in place until discharge from the recovery room. All patients will have CBC drawn on post operative day 1, as is the standard of care at our institution. Based on the drop in hemoglobin from pre-op to post-op day 1, patients will be separated into quartiles. The quartile with the highest drop in hemoglobin will be the "cases" and compared to the remainder of the quartiles or "controls." In addition, values obtained from the non-invasive monitor will be compared to those obtained from CBC.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing primary cesarean delivery after failed induction of labor, or repeat cesarean delivery after failed TOLAC (trial of labor after cesarean)
* Pregnant women between the ages of 18-50

Exclusion Criteria:

* Patient who are not pregnant
* Patients unwilling or unable to provide consent
* Patients under the age of 18
* Patients who are incarcerated

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine H Jelliffe, MD, Principal Investigator — University of Texas; Antonio F Saad, MD, Study Director — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 65
Age, Continuous [Mean (Full Range); unit: years] | 26.9 [19 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 11
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Pearson Correlation Coefficient for Hemoglobin Measurements
Description: Pearson Correlation Coefficient for hemoglobin measurements (Difference in Hemoglobin blood counts in g/dL between preop and post operative levels) obtained from blood draw to those obtained from the monitor
Time Frame: 1 day post partum
Population: This value was compared to post operative day 1 hemoglobin from a complete blood count testing. We used Pearson correlation analysis.
  range of values from +1 to -1. A value of 0 indicates that there is no association between the two variables. A value greater than 0 indicates a positive association;
Measure: Number; unit: Correlation Coeficient
Groups:
- End of Case Non-invasive Hemogblobin: This value was obtained from the non-invasive device at the end of the case (hemoglobin g/dL).
Arm/Group | End of Case Non-invasive Hemogblobin
Number analyzed (Participants) | 19
Correlation Coeficient | 0.6

2. Secondary Outcome: Number of Participants Who Required Blood Transfusion
Description: The rates in percentage of patients that received transfusion of packed red blood cells.
Time Frame: 0-5 days post partum
Population: Among all participant, the ncount of participants that received blood transfusion.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 65
Participants | 65

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT03150043/Prot_SAP_000.pdf